CLINICAL TRIAL: NCT06376617
Title: Pattern Of Isolated Fungi From Bronchoalveolar Lavage Among Patients With Bronchial Asthma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Tamer Awad, lecturer of chest medicine, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MS.24.03.2743
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Bronchial Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: BAL will stained by fungal staining with lactophenol stain as well as culture on Sabouraud dextrose agar.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study patern of fungal inection which cause excerbation (Other): Take bal through fob and send for fungal stain and culure
  Interventions: Device: fibroptic bronchoscopy

INTERVENTIONS:
Device: fibroptic bronchoscopy — take bal through fibrooptic bronchoscopy and send for stain and culcure
  Other Names: fugnal stain and culcure

SUMMARY:
This study is to assess the pattern of isolated fungi from the respiratory air way (bronchial tree) from bronchoalvealar lavage (BAL) in asthmatic patients with uncontrolled or difficult to treat asthma

DETAILED DESCRIPTION:
Asthma is a heterogeneous disease, usually characterized by chronic airway inflammation and hyper responsiveness. It is defined by the history of respiratory symptoms, such as wheeze, shortness of breath, chest tightness and cough, that vary over time and in intensity, together with variable expiratory airflow limitation. Airflow limitation may later become persistent Making the diagnosis of asthma is based on identifying both a characteristic pattern of respiratory symptoms such as wheezing, shortness of breath (dyspnea), chest tightness or cough, and variable expiratory airflow limitation (Levy ML et al,2006 ) In asthma, lung function may vary between completely normal and severely obstructed in the same patient. Poorly controlled asthma is associated with greater variability in lung function than well-controlled asthma (Graham BL et al,2019 ) A reduced FEV1 may be found with many other lung diseases (or poor spirometric technique), but a reduced ratio of FEV1 to forced vital capacity (FEV1/FVC), compared with the lower limit of normal, indicates expiratory airflow limitation Most patients with asthma can be well-controlled with low doses of anti- inflammatory agents. However, up to 10% of patients with asthma manifest with severe disease, which leads to considerable limitation of activities of daily life and can be fatal .(Moore et al.,2007).

Severe asthma remains a challenge for patients and clinicians, as these patients are not only difficult to treat but also contribute disproportionately to the overall costs of asthma .

The reasons for the variation in severity of asthma from patient to patient are not fully understood. Several environmental factors, such as house dust mite, animal dander from pets, and environmental fungi (especially their continued exposure), are known to worsen asthma control (GINA ,2023).

Fungal diseases are a concern in the medical and public health community because of the increasing number of people with weakened immune systems and the advances in health care practices.

Fungi can be linked to severe asthma in a multitude of ways, including (inhalation of fungal spores; fungal sensitization,and allergic bronchopulmonary aspergillosis (ABPA) a severe degree of fungal sensitization culminating in irreversible bronchopulmonary damage Fungal infections are difficult to diagnose because clinical symptoms, signs, and radiographic manifestations are unspecific. Therefore, a definitive diagnosis requires direct identification of fungi from the site of infection.

Funal infection of air way can be diagnosed by :

* Microscopic Examination
* Culture of respiratory secretions (sputum,BAL), tissue samples, or blood.
* Serology : assay of serum that detect host antibodies reacting to fungal elements.
* Antigen antibodie :detection of components of the fungal wall that are shed into the bloodstream or other body fluids as the organism proliferates.
* PCR Up to 70% of severe asthmatics are IgE sensitized to fungi compared with 10% of mild-to-moderate asthmatics and 5% of the general population (RICK et al.,2020).

Exposure to outdoor fungal spores has been associated with worsening asthma symptoms, poor lung function, hospital admissions, and asthma- related death.(Agarwal et al.,2011).

Bronchoscopy is used as a diagnostic tool to observe endobronchial lesions and to obtain clinical specimens such as bronchoalveolar lavage (BAL) and bronchial washing. Fungal culture examination from clinical specimen of bronchoscopy could assist in diagnosing pulmonary mycosis (Hermansyah et al.,2021).

Bronchoalveolar lavage (BAL) is a common and relatively safe diagnostic procedure for the evaluation of patients with lung disease. It often provides valuable diagnostic information when clinical history, physical exam, routine laboratory testing, pulmonary function testing and radiographic imaging are insufficient to reach a definitive diagnosis. Compared to sputum analysis, BAL allows for targeted sampling of the lower respiratory tract with less microbial contamination from the upper aerodigestive tract (Davidson et al.,2020).

Aim of Work:

The aim of this study is to assess the pattern of isolated fungi from the respiratory air way (bronchial tree) from bronchoalvealar lavage (BAL) in asthmatic patients with uncontrolled or difficult to treat asthma .

Study Design:

Prospective, cross sectional, observational study . study locality: All adult patients (>18 years) with difficult to treat bronchial asthma or frequent exacerbation , admitted to or follow in outpatient clinic in Mansoura University chest department and Damietta chest hospital .

Sample Size :

(BAL) will collected from 60 patients with bronchial asthma

Patients and Methods:

Patients with Uncontrolled bronchial asthma, frequent exacerbations and difficult to treat symptoms despite adherence to medication according to (GINA 2023).

Patients will classified according to Asthma Control Questionnaire (ACQ GINA2023 Asthma Control Questionnaire (ACQ):

In the past 4 weeks, has the patient had:

* Daytime asthma symptoms more than twice/week? Yes No
* Any night waking due to asthma? Yes No
* SABA* reliever for symptoms more than twice/week? Yes No
* Any activity limitation due to asthma? Yes NO Well controlled: Non of these . Partly controlled: 1-2 Uncontrolled :3-4 Inclusion criteria

  * Age 18 years or more.
  * Patients with Uncontrolled bronchial asthma, frequent exacerbations and difficult to treat symptoms despite adherence to medication.

Exclusion criteria

1. Age less than 18 years.
2. Patients who do not give consent for the procedure.
3. Patients with unstable cardiac conditions (recent myocardial infarction, cardiac arrhythmia, etc.)
4. Pregnant women.
5. Patient already on antifungal treatment.
6. Bleeding profile abnormality.
7. patients during acute sever attacks .

All the patients will be subjected to the following:

1. Clinical evaluation:

   - Full history taking and clinical examination.
2. Laboratory work up:

   * CBC
   * Bleeding profile (INR)
3. ECG
4. pulmonary function test (pfts)with reversibility test Positive bronchodilator (BD) responsiveness (reversibility test) Is consider in adults if : increase in FEV1 of >12% and >200 mL (greater confidence if increase is >15% and >400 mL).

Measure change 10-15 minutes after 200-400 mcg salbutamol (albuterol) or equivalent, compared with pre-BD readings.

Before bronchodilator reversibility testing, short-acting and long-acting inhaled bronchodilators were withheld 4 and 12 hours; short-acting and long-acting oral bronchodilators were withheld 8 and 12 hours before testing, respectively Radiological work up

- CT chest or chest x ray 6- Bronchoscopy with BAL: Bronchoscopy with BAL was performed according to standardized procedures designed to minimize oral contamination. BAL was performed by sequentially instilling and then withdrawing 50 ml aliquots of sterile normal saline.

Bronchoalveolar lavage fluid specimens collected under aseptic precautions was immediately transported to the laboratory for fungal processing BAL fluid should be collected in a labeled sterile container and transported expediently to the laboratory for analysis.

Microbiology work up :

BAL will stained by fungal staining with lactophenol stain as well as culture on Sabouraud dextrose agar.

Some pathogenic fungi grow slowly in culture and require plates to be held for up to 2 weeks, and in some case up to 4 weeks, before being discarded as negative. However, many common pathogenic fungi, such as Aspergillus fumigatus and Candida albicans, will produce identifiable colonies within 1-3days. Cultures should be examined at frequent intervals (at least three times weekly) .

Statistical analysis:

The collected data will be coded, processed and analyzed using SPSS program (Version 26) for windows. The appropriate statistical tests will be used when needed. P values less than 0.05 (5%) will be considered to be statically significant.

Ethical consideration:

* Study protocol will be submitted for approval by IRB
* Approval of the mangers of the health care facilities in which the study will be conducted
* Informed written consent will be obtained from each participant sharing in the study.
* Confidentiality and personal privacy will be respected in all levels of the study. Collected data will not be used for any other purpose

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or more.
2. Patients with Uncontrolled bronchial asthma, frequent exacerbations and difficult to treat symptoms despite adherence to medication.

Exclusion Criteria:

1. Age less than 18 years.
2. Patients who do not give consent for the procedure.
3. Patients with unstable cardiac conditions (recent myocardial infarction, cardiac arrhythmia, etc.)
4. Pregnant women.
5. Patient already on antifungal treatment.
6. Bleeding profile abnormality.
7. patients during acute sever attacks .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-25 (Estimated); Primary Completion 2025-04-20 (Estimated); Study Completion 2025-05-20 (Estimated)

PRIMARY OUTCOMES:
assess the pattern of isolated fungi from the respiratory air way (bronchial tree) from bronchoalvealar lavage (BAL) in asthmatic patients with uncontrolled or difficult to treat asthma | 1 year
  BAL will stained by fungal staining with lactophenol stain as well as culture on Sabouraud dextrose agar.